CLINICAL TRIAL: NCT03880617
Title: Yeur-Hur Lai, PhD, RN, School of Nursing, College of Medicine, National Taiwan University
Brief Title: Distress, Medication Adherence and Care Needs in Patients With CML and GIST Receiving Oral Targeted Therapy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201501004RIND
Record Dates: First submitted 2018-12-03; First posted 2019-03-19 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2019-12

CONDITIONS: CML; GIST
Keywords: Chronic myeloid leukemia; Gastrointestinal stromal tumor; Targeted therapy; Care needs; Medication adherence
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Myeloid Leukemia (CML): For CML, the first-line targeted drug is imatinib, and then second line as nilotinib and dasatinib. In the past, the median survival of CML is around 4 to 6 years (NCI, 2008). Fortunately, the launch of the targeted therapy, the median survival is expected to approach normal life expectancy for most patients. However, limited to the less than 20 years of advent of TKI, the exact effects on survival time is not yet determined.
- Gastrointestinal Stromal Tumor (GIST): For patients with GIST, the imatinib mesylate (Glivec, Novartis Pharma, Basel, Switzerland) (Heinrich et al, 2003) is the first line drug and sunitinib as the second line drug. Sunitinib is an anti-angiogenesis agent by virtue of targeting multiple tyrosine kinases, including the vascular endothelial growth factor receptors (VEGFR). With these target drugs, the survival of advanced GIST patients is prominently prolonged (Lamba, Ambrale, Lee, Gupta, Rafiyath, & Liu D, 2012). The median overall survival (OS) of advanced GIST patients increased from 18 to 57 months with imatinib therapy (Blanke et al, 2008).

SUMMARY:
Background: Long-term or life-long oral targeted therapy might also increase patients' distress, influencing patients' cognitive and life activity function, medication adherence and related care needs. However, very limited information has been known about patients' experiences.

Purpose: First, to examine the changes of perceived physical and psychological distress, functional status, medication adherence, and unmet care needs; and second, to identify factors related to the changes of patients' medication adherence and unmet care needs by generalized estimating equation (GEE).

Methods: This is a two-phase study. Phase I is a cross-sectional survey study, and the second phase is a 1-year follow-up prospective longitudinal study. Eligible subjects are CML and GIST patients newly taking oral targeted therapy. Patients will be assessed before taking the first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively). The patients were assessed of their (1) symptom severity, (2) psychological distress, (3) cognitive and life activity function, (4) adherence, (5) social support, (6) unmet care needs, and (7) background and disease-treatment information. Data will be analyzed mainly by GEE to identify the predictors (independent variables) of the changes in medication adherence and unmet care needs overall the 12 months, 6 time points. After the approval of IRB, research assistants in different data collection sites will be trained for maintaining the consistency and quality of data collection.

Expected Outcomes and Future Implications: Although CML and GIST are not the most prevalent cancers in Taiwan, the investigators aim to use both groups of patients groups to examine the current status and changes of distress, adherence and care needs in patients are taking long-term or life-long TKI derived oral targeted therapy. From Phase II study, the changes of newly TKI targeted therapy takers' distress, adherence and care needs would be carefully and in-depth examined. It will provide health care professionals a more comprehensive picture of the changes in patients' distress, adherence, and care needs during taking oral targeted therapy. The results will also provide as a basis and evidence for better development a timing and comprehensive care models to fit and increase patients' life quality during receiving the most advanced targeted therapy.

DETAILED DESCRIPTION:
Prospective Panel Study, a 12-month follow-up longitudinal study. Eligible subjects are newly diagnosed CML and GIST patients who need to take targeted therapy. Patients would be assessed on the time point of before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively). Before this study conducted, the institutional review board would review the study. The research nurses will approach potential participants after their patients were initial treating oral targeted therapy and invite them to enroll in the study. Potential participants would be informed of the study purposes and interview contents. After written consent is obtained, the interview will be arranged. In order to control the quality of data collection, the investigators will train these research assistants. Research training will include ethical concerns about the collection of research data, methods of approaching eligible subjects, interviewing techniques, and pilot testing of data collection. The training will provide research assistants by the PI and Co-PI of this study. Training for research assistants.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed CML and GIST patients
* patients need to take targeted therapy

Exclusion Criteria:

* conscious unclear
* recurrence or with bone meta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion criteria was (1) adults diagnosed with CML or GIST; (2) awareness of their diagnosis; (3) who are new user of targeted therapy and before their first dosage; and (4) agree to participate in the study after its purposes and procedures have been explained. Exclusion criteria was: (1) Patients with CML did not have targeted therapy currently or who are receiving chemotherapy; and (2) GIST patients who only received surgery; or who did not receive targeted therapy currently. Consecutive patients will be approached and recruited from both hematological and gastroenterological OPD at a medical center in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity Scale (SSS) | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  The 43-item Symptom Severity Scale (SSS) was modified from the Symptom Distress Scale (SDS) (McCorkle & Young, 1978). The SSS aims to assess the level of symptom severity with Each item scored from 0 to 10 (0 = do not have the problem at all, 10 = the most severity that I have ever experienced). The higher the score indicated the higher the symptom severity. The SSS has been used in the previous study and had good reliability and validity (Chen, Liao, Lin, Chang, & Lai, 2009; Lai et al., 2003; Shun et al., 2008).
Change in Hospital Anxiety and Depression Scale (HADS) - Depression Subscale | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  We will use 14-item HADS to assess patients' anxiety and depression (Zigmond & Snaith, 1983). The HADS has 7 items that measure anxiety and 7 that measure depression. The total score of each subscale is ranged from 0 to 21 with a higher score indicating a higher level of anxiety and depression. The Taiwanese version of HADS has been developed and validated showed promising psychometrics (Chen et al., 2010; Cheng, Hao, Lin, & Yeh, 2000).
Change in Fear of Cancer Recurrence Index-42 (FCRI-42) | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  The 42-item FCRI will be used to measure patients' self-reported fear of cancer recurrence (Simard & Savard, 2009) and it currently has been applied to several kinds of cancer populations (Simard & Savard, 2009). FCRI measures seven dimensions of fear of cancer recurrence. It is a five-point Likert's scale (0-4 for each item, scoring from 0 to 168 for total scale) and generally with higher scores indicates higher fear of recurrence. The Chinese version has been translated and validated in PI's on-going early-stage lung cancer study and proved to be psychometrically satisfied.
Change in WHO Disability Assessment Schedule 2.0 (WHO DAS 2.0) - Cognition and Life Activity Subscales | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  WHODAS 2.0 has been developed based on the International Classification of Functioning, Disability, and Health (ICF) published by the World Health Organization (WHO) in 2001. In this study, we particularly apply the 6-item cognition subscale which to assess a person's cognition and thinking abilities. In addition, the 8-item life activities subscale will assess changes in life activities after having cancer and taking targeted therapy. Each scale of subscale was standardized from 0 to 100, with a higher score indicating higher limitation in daily life. The Chinese version has been tested of its psychometrics in chronic illness patients and found to be reliable (Chi et al., 2014; Chiu et al., 2014; Yen et al., 2014).
Change in Medical Outcome Study Social Support Survey (MOS-SSS) - Short form | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  We will use the MOS-SSS to assess patient perceived social support (Sherbourne & Stewart, 1991). The 20-item MOS-SSS consists of four subscales: emotional/informational support (8 items), tangible support (4 items), affectionate 11 support (3 items), and positive social interaction (3 items), and additional item (I item). The score for each item ranges from 1 (not at all) to 5 (very much). The summed scores of each domain and the global scale are converted into standardized scores ranging from 0 to 100, with higher scores representing more support. Several previous studies have demonstrated satisfactory psychometric characteristics for this scale (Moser, Stuck, Silliman, Ganz, Clough-Gorr, 2012; Yu, Lee, Woo, 2004).
Change in Supportive Care Needs Survey (SCNS-9) | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  The brief version of SCNS-ST9 includes 9 items identified from SCNS-34. Each item with the following response options: "No need, not applicable (1)"; "No need, satisfied (2)"; "Low need (3)"; "Moderate need (4)"; "High need (5)". The number of items with moderate/high needs was counted for each domain of the SCNS-9 and the sum of item scores was transformed to a standardized score (0-100) with higher scores indicating more unmet needs. The SCNS-ST9 had good validity and reliability (Boyes, Girgis, & Lecathelinais, 2009; Girgis, Stojanovski, Boyes, King, & Lecathelinais, 2012).
Change in Background, Disease and Treatment Information Form (BDTIF) | Patients will be assessed before taking first targeted therapy and 1st, 2nd, 3rd, 6th, 12th month (T1-T6, respectively)
  In addition to patients' demographic information (age, gender, education). Disease and treatment-related variables include: (1) types of diagnosis, (2) Performance status (by Karnofsky Performance Index), (3) length of time diagnosis (month), (4) Duration of receiving targeted therapy (months), (5) types of targeted therapy, (6) Dosages of target therapy, (7) Times of medication taking per day, and (8) Time since cancer diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hosptial, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Lamba G, Ambrale S, Lee B, Gupta R, Rafiyath SM, Liu D. Recent advances and novel agents for gastrointestinal stromal tumor (GIST). J Hematol Oncol. 2012 May 8;5:21. doi: 10.1186/1756-8722-5-21. PMID 22569033
- [Background] Blanke CD, Rankin C, Demetri GD, Ryan CW, von Mehren M, Benjamin RS, Raymond AK, Bramwell VH, Baker LH, Maki RG, Tanaka M, Hecht JR, Heinrich MC, Fletcher CD, Crowley JJ, Borden EC. Phase III randomized, intergroup trial assessing imatinib mesylate at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumors expressing the kit receptor tyrosine kinase: S0033. J Clin Oncol. 2008 Feb 1;26(4):626-32. doi: 10.1200/JCO.2007.13.4452. PMID 18235122
- [Background] McCorkle R, Young K. Development of a symptom distress scale. Cancer Nurs. 1978 Oct;1(5):373-8. No abstract available. PMID 250445
- [Background] Lai YH, Chang JT, Keefe FJ, Chiou CF, Chen SC, Feng SC, Dou SJ, Liao MN. Symptom distress, catastrophic thinking, and hope in nasopharyngeal carcinoma patients. Cancer Nurs. 2003 Dec;26(6):485-93. doi: 10.1097/00002820-200312000-00008. PMID 15022980
- [Background] Chen SC, Liao CT, Lin CC, Chang JT, Lai YH. Distress and care needs in newly diagnosed oral cavity cancer patients receiving surgery. Oral Oncol. 2009 Sep;45(9):815-20. doi: 10.1016/j.oraloncology.2009.01.001. Epub 2009 Feb 27. PMID 19250858
- [Background] Shun SC, Chiou JF, Lai YH, Yu PJ, Wei LL, Tsai JT, Kao CY, Hsiao YL. Changes in quality of life and its related factors in liver cancer patients receiving stereotactic radiation therapy. Support Care Cancer. 2008 Sep;16(9):1059-65. doi: 10.1007/s00520-007-0384-y. Epub 2008 Jan 16. PMID 18197433
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Lampic C, von Essen L, Peterson VW, Larsson G, Sjoden PO. Anxiety and depression in hospitalized patients with cancer: agreement in patient-staff dyads. Cancer Nurs. 1996 Dec;19(6):419-28. doi: 10.1097/00002820-199612000-00002. PMID 8972974
- [Background] Chen SC, Lai YH, Liao CT, Lin CC, Chang JT. Changes of symptoms and depression in oral cavity cancer patients receiving radiation therapy. Oral Oncol. 2010 Jul;46(7):509-13. doi: 10.1016/j.oraloncology.2010.02.024. Epub 2010 Mar 21. PMID 20308004
- [Background] Cheng PT, Hao SP, Lin YH, Yeh AR. Objective comparison of shoulder dysfunction after three neck dissection techniques. Ann Otol Rhinol Laryngol. 2000 Aug;109(8 Pt 1):761-6. doi: 10.1177/000348940010900811. PMID 10961810
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Simard S, Savard J. Screening and comorbidity of clinical levels of fear of cancer recurrence. J Cancer Surviv. 2015 Sep;9(3):481-91. doi: 10.1007/s11764-015-0424-4. Epub 2015 Jan 21. PMID 25603948
- [Background] Chi WC, Chang KH, Escorpizo R, Yen CF, Liao HF, Chang FH, Chiou HY, Teng SW, Chiu WT, Liou TH. Measuring disability and its predicting factors in a large database in Taiwan using the World Health Organization Disability Assessment Schedule 2.0. Int J Environ Res Public Health. 2014 Nov 25;11(12):12148-61. doi: 10.3390/ijerph111212148. PMID 25429682
- [Background] Chiu TY, Yen CF, Chou CH, Lin JD, Hwang AW, Liao HF, Chi WC. Development of traditional Chinese version of World Health Organization disability assessment schedule 2.0 36--item (WHODAS 2.0) in Taiwan: validity and reliability analyses. Res Dev Disabil. 2014 Nov;35(11):2812-20. doi: 10.1016/j.ridd.2014.07.009. Epub 2014 Aug 3. PMID 25094056
- [Background] Yen CF, Hwang AW, Liou TH, Chiu TY, Hsu HY, Chi WC, Wu TF, Chang BS, Lu SJ, Liao HF, Teng SW, Chiu WT. Validity and reliability of the Functioning Disability Evaluation Scale-Adult Version based on the WHODAS 2.0--36 items. J Formos Med Assoc. 2014 Nov;113(11):839-49. doi: 10.1016/j.jfma.2014.08.008. Epub 2014 Oct 5. PMID 25294100
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Moser A, Stuck AE, Silliman RA, Ganz PA, Clough-Gorr KM. The eight-item modified Medical Outcomes Study Social Support Survey: psychometric evaluation showed excellent performance. J Clin Epidemiol. 2012 Oct;65(10):1107-16. doi: 10.1016/j.jclinepi.2012.04.007. Epub 2012 Jul 20. PMID 22818947
- [Background] Yu DS, Lee DT, Woo J. Psychometric testing of the Chinese version of the medical outcomes study social support survey (MOS-SSS-C). Res Nurs Health. 2004 Apr;27(2):135-43. doi: 10.1002/nur.20008. PMID 15042639
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Kekale M, Talvensaari K, Koskenvesa P, Porkka K, Airaksinen M. Chronic myeloid leukemia patients' adherence to peroral tyrosine kinase inhibitors compared with adherence as estimated by their physicians. Patient Prefer Adherence. 2014 Nov 24;8:1619-27. doi: 10.2147/PPA.S70712. eCollection 2014. PMID 25473270
- [Background] Khosravizade Tabasi H, Madarshahian F, Khoshniat Nikoo M, Hassanabadi M, Mahmoudirad G. Impact of family support improvement behaviors on anti diabetic medication adherence and cognition in type 2 diabetic patients. J Diabetes Metab Disord. 2014 Nov 25;13(1):113. doi: 10.1186/s40200-014-0113-2. eCollection 2014. PMID 25436202
- [Background] Boyes A, Girgis A, Lecathelinais C. Brief assessment of adult cancer patients' perceived needs: development and validation of the 34-item Supportive Care Needs Survey (SCNS-SF34). J Eval Clin Pract. 2009 Aug;15(4):602-6. doi: 10.1111/j.1365-2753.2008.01057.x. Epub 2009 Jun 10. PMID 19522727
- [Background] Girgis A, Stojanovski E, Boyes A, King M, Lecathelinais C. The next generation of the supportive care needs survey: a brief screening tool for administration in the clinical oncology setting. Psychooncology. 2012 Aug;21(8):827-35. doi: 10.1002/pon.1973. Epub 2011 Apr 12. PMID 21484938
- See also: National Cancer Institute (2008). Cancer Stat Facts: Leukemia - Chronic Myeloid Leukemia (CML). — https://seer.cancer.gov/statfacts/html/cmyl.html